CLINICAL TRIAL: NCT03582124
Title: A Phase I/II Study Evaluating the Safety and Pharmacokinetics of Panitumumab-IRDye800 as an Optical Imaging Agent to Detect Lung Cancer During Surgical Procedures
Brief Title: Panitumumab-IRDye800 in Detecting Cancer in Participants With Lung Cancer During Surgery
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-41302; NCI-2018-00494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0099 (Other: OnCore)
Record Dates: First submitted 2018-06-14; First posted 2018-07-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Carcinoma; Metastatic Malignant Neoplasm in the Lung; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (panitumumab-IRDye800, surgery, NIR) (Experimental): Participants receive panitumumab- IRDye800 IV over 60 minutes on day 0, and then undergo NIR and surgery within 1-5 days.
  Interventions: Procedure: Near-Infrared Fluorescence Imaging; Drug: Panitumumab-IRDye800; Other: Pharmacokinetic Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Near-Infrared Fluorescence Imaging — Undergo imaging
  Other Names: NIR Fluorescence Imaging; NIR Optical Imaging
Drug: Panitumumab-IRDye800 — Given IV
  Other Names: Panitumumab IRDye 800; RDye800-Panitumumab Conjugate
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase I/II trial studies the best dose and timing of panitumumab-IRDye800 in detecting cancer in participants with lung cancer during the surgery. Panitumumab-IRDye800 is a combination of the antibody drug panitumumab and IRDye800CW, an investigational dye that can be seen using a special camera. Panitumumab-IRDye800 may attach to tumor cells and make them more visible during surgery in patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the optimal dose and timing of panitumumab IRDye800 infusion for identifying lung cancer compared to surrounding normal tissue in the ex vivo setting as measured by tumor to background ratio.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of the panitumumab IRDye800 as an imaging agent in subjects undergoing resection of lung cancer.

II. Determine whether the primary lung tumor or positive lymph nodes can be detected by near-infrared (NIR) fluorescence imaging with panitumumab IRDye800 but not by white light imaging.

OUTLINE: This is a phase I, dose-escalation study of panitumumab-IRDye800 followed by a phase II study.

Participants receive panitumumab- IRDye800 intravenously (IV) over 60 minutes on day 0, and then undergo NIR and surgery within 1-5 days.

After completion of study treatment, participants are followed up for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung nodule or mass concerning for malignancy, either primary lung cancer or lung metastases, whether or not it is biopsy-proven
* Patients scheduled to undergo planned standard of care surgical resection for a lung nodule or mass with diagnostic and/or curative intent for lung cancer
* Karnofsky performance status of at least 70% or Eastern Cooperative Oncology Group (ECOG)/Zubrod level 0-2
* Hemoglobin ≥ 9 gm/dL
* White blood cell count > 3000/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 1.5 times upper reference range

Exclusion Criteria:

* Received an investigational drug within 30 days prior to first dose of panitumumab-IRDye800
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* History of infusion reactions to monoclonal antibody therapies
* Pregnant or breastfeeding
* Magnesium or potassium lower than the normal institutional values
* Subjects receiving class IA (quinidine, procanamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* Prisoners, institutionalized individuals, and patients unable to consent for themselves

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Tumor to background ratio (TBR), measured in ex vivo tissues | Up to 1 year
  The TBR is defined as the near-infrared fluorescence signal of tumor or lymph node tissue compared to normal adjacent tissue measured in ex vivo tissues. Outcomes will be reported as the TBR (mean) and standard deviation for each dose group and timing group (1-2 days or 3-5 days prior to surgery).

SECONDARY OUTCOMES:
Number of Grade 2 or higher AEs determined to be clinically significant and definitely, probably or possibly related to study drug | Up to 30 days
Metastatic lesion detection by Panitumumab-IRDye800 versus standard assessments | Up to 1 year
  Intraoperative near-infrared fluorescence imaging with panitumumab-IRDye800 will be compared to conventional white light visualization and ex vivo histopathology methods to identify metastatic lesions. Outcomes will be reported as the number of metastatic lesions detected by both near-infrared fluorescence imaging and histopathology, and each method alone.
Tumor-positive lymph node detection by Panitumumab-IRDye800 versus standard assessments | Up to 1 year
  Intraoperative near-infrared fluorescence imaging with panitumumab-IRDye800 will be compared to conventional white light visualization and ex vivo histopathology methods to identify tumor-positive lymph nodes. Outcomes will be reported as the number of tumor-positive lymph nodes detected by both near-infrared fluorescence imaging and histopathology, and each method alone.
Residual disease detection by Panitumumab-IRDye800 versus standard assessments | Up to 1 year
  Intraoperative near-infrared fluorescence imaging with panitumumab-IRDye800 will be compared to conventional white light visualization and ex vivo histopathology methods to identify residual disease at resection margins. Outcomes will be reported as the number of positive-margins detected by both near-infrared fluorescence imaging and histopathology, and each method alone.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Lui, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States